CLINICAL TRIAL: NCT03181685
Title: Subcutaneous Versus Vaginal Progesterone as Luteal Support in IVF/ICSI Cycles: Which is the Preference Expressed by the Patients?
Brief Title: Patients' Preference for Subcutaneous or Vaginal Progesterone as Luteal Support in IVF/ICSI Cycles
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: 27 couples were recruited. This unexpected poor recruitment was due to more clinical pregnancies (for a better patients' selection) and more freeze-all cycles.
Sponsor: Andros Day Surgery Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Andros Day Surgery Clinic
Record Dates: First submitted 2017-05-31; First posted 2017-06-09 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Infertility; In Vitro Fertilization
Keywords: Progesterone supplementation; IVF; Preference expressed by the patient
MeSH Terms: conditions — Infertility | interventions — Progesterone; Injections, Subcutaneous; follitropin alfa; cetrorelix

STUDY DESIGN:
Intervention Model Description: This is randomized, controlled, prospective, crossover, open-label, two-treatments, two-period trial
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment S (Subcutaneous) (Active Comparator): Progesterone 25 mg subcutaneous (a single administration per day) from the day of oocyte retrieval. Controlled ovarian stimulation (COS) will be performed with recombinant FSH and cetrorelix acetate.
  Interventions: Drug: Progesterone 25 MG subcutaneous; Drug: recombinant FSH; Drug: Cetrorelix Acetate
- Treatment V (Vaginal) (Active Comparator): Micronized progesterone 200 mg (3 vaginal administrations per day) from the day of oocyte retrieval. Controlled ovarian stimulation (COS) will be performed with recombinant FSH and cetrorelix acetate.
  Interventions: Drug: Micronized progesterone 200 MG; Drug: recombinant FSH; Drug: Cetrorelix Acetate

INTERVENTIONS:
Drug: Progesterone 25 MG subcutaneous — A single subcutaneous administration per day from the day of oocyte retrieval
  Other Names: Pleyris
  Arms: Treatment S (Subcutaneous)
Drug: Micronized progesterone 200 MG — 3 vaginal administrations per day from the day of oocyte retrieval
  Other Names: Prometrium
  Arms: Treatment V (Vaginal)
Drug: recombinant FSH — Controlled ovarian stimulation (COS)
  Other Names: Gonal-f
Drug: Cetrorelix Acetate — Inhibition of Luteinizing Hormone (LH) premature surge during COS
  Other Names: Cetrotide

SUMMARY:
This randomized, controlled, prospective, crossover, open-label, two-treatments, two-period trial aimed to evaluate the preference expressed by the patient concerning the subcutaneous administration of progesterone versus the vaginal one.

The couples, scheduled for performing 2 In Vitro Fertilization (IVF)/Intracytoplasmic Sperm Injection (ICSI) cycles will be randomized to receive, as luteal phase supplementation, Pleyris 25 milligram (mg) (a single subcutaneous administration per day) or Prometrium 200 mg (3 vaginal administrations per day).

DETAILED DESCRIPTION:
Each participant will receive both treatments. During the first IVF/ICSI cycle, the luteal phase will be supplemented with subcutaneous progesterone (S) or vaginal progesterone (V). At the end of the cycle (on the day of beta-hCG), a survey for determining the level of satisfaction will be administered and filled in by the patient during the waiting time and always before the knowledge of the result. This practical organization allows the elimination of emotional biases correlated with the outcome. In case of a negative beta-hCG, the patient will be scheduled for a second IVF/ICSI cycle after a washout (W) period (between 2 and 6 months). In the second cycle, the patient will undergo, during the luteal phase, the opposite treatment (V or S). Also in this case, the survey for evaluating the level of satisfaction will be administered on the day of beta-hCG, with the same modalities of the first cycle. The domains of the surveys are focused on facility of the administration, comfort, level of complaint, side effects, overall level of satisfaction.

The sequence S-V or V-S will be randomly assigned (random assignment) with the concealment of the allocation.

In case of a negative beta-hCG also in the second cycle, a post-hoc comparison between the two treatments will be carried out through a Semantic Differential Scale, in the "follow-up" phase.

ELIGIBILITY:
Inclusion Criteria:

first IVF/ICSI attempt (at the enrolment), regular menstrual cycles (25-33 days), controlled ovarian stimulation performed with Gonadotropin Releasing Hormone (GnRH) antagonists and gonadotrophins (recombinant FSH)

Exclusion Criteria:

systemic diseases, chronic medical therapies, pregnancy in one of the IVF/ICSI cycles, embryo "freeze all" strategy in one of the IVF/ICSI cycles for preventing Ovarian Hyperstimulation Syndrome (OHSS)

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Surveys for testing the satisfaction | Single administration at the end of each treatment cycle (an average of 28 days)
  Patient's level of satisfaction will be measured as score on 5-point likert scale + 2 qualitative response

SECONDARY OUTCOMES:
Semantic Differential Scale | Single administration at the end of two treatment cycles (an average of 130 days)
  Patient's preference of treatment measured on a 7-point likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Allegra, MD, Principal Investigator — Andros Day Surgery Clinic
Locations (1):
- ANDROS Day Surgery Clinic, Reproductive Medicine Unit, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beltsos AN, Sanchez MD, Doody KJ, Bush MR, Domar AD, Collins MG. Patients' administration preferences: progesterone vaginal insert (Endometrin(R)) compared to intramuscular progesterone for Luteal phase support. Reprod Health. 2014 Nov 11;11:78. doi: 10.1186/1742-4755-11-78. PMID 25385669
- [Background] van der Linden M, Buckingham K, Farquhar C, Kremer JA, Metwally M. Luteal phase support for assisted reproduction cycles. Cochrane Database Syst Rev. 2015 Jul 7;2015(7):CD009154. doi: 10.1002/14651858.CD009154.pub3. PMID 26148507
- [Background] Yanushpolsky E, Hurwitz S, Greenberg L, Racowsky C, Hornstein M. Crinone vaginal gel is equally effective and better tolerated than intramuscular progesterone for luteal phase support in in vitro fertilization-embryo transfer cycles: a prospective randomized study. Fertil Steril. 2010 Dec;94(7):2596-9. doi: 10.1016/j.fertnstert.2010.02.033. Epub 2010 Mar 27. PMID 20347079